CLINICAL TRIAL: NCT01060059
Title: EBIRIOS - Exenatide and Basal Insulins Use in the Real Setting: an Italian Observational Study in Patients With Type 2 Diabetes and Secondary Failure of Oral Antihyperglycemic Treatment
Brief Title: Exenatide and Basal Insulins Use in the Real Setting: an Observational Study in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: H8O-IT-B014
Record Dates: First submitted 2010-01-26; First posted 2010-02-02 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Byetta; basal insulin; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exenatide: The targeted population consists of adult patients with type 2 Diabetes Mellitus unable to achieve the desired level of glycemic control while using oral anti-hyperglycemic agents and who initiate treatment with exenatide.
  Interventions: Drug: exenatide
- basal insulin: The targeted population consists of adult patients with type 2 Diabetes Mellitus unable to achieve the desired level of glycemic control while using oral anti-hyperglycemic agents and who initiate treatment with basal insulin.
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: BYETTA
  Groups: exenatide
Drug: basal insulin — subcutaneous injection, dosing according to physician's clinical judgment
  Groups: basal insulin

SUMMARY:
Although the efficacy and safety profile of exenatide has been well established, few data exist on the real world results of exenatide treatment in specific populations and clinical settings. This study is intended to fill this gap through observing and collecting prospective data from a population of Italian patients initiating treatment with either exenatide or basal insulin formulations after failure to achieve glycemic control with oral antihyperglycemic agents (OHA).

Observational studies represent noninterventional research; therefore, this study does not involve randomization of patients to particular comparator arms or therapies. The term "noninterventional" means that the healthcare providers decisions regarding the proper treatment and care of the patient are made in the course of normal clinical practice. Patients enrolled in this study are enrolling for the collection of their data on observations made during normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Are inadequately controlled with single or multiple OHA as evidenced by an HbA1c > 7.0%
2. Have presented during the routine course of care and, together with their physician, have decided to initiate treatment with either exenatide twice daily or conventional insulin therapy with basal insulin (insulin glargine, detemir, protaminated insulin lispro, protaminated human insulin) added to the existing treatment with OHA
3. Have not been treated with GLP-1 receptor agonist for more than 7 consecutive days within 3 months before entering the study
4. Have not been treated with insulins for more than 7 consecutive days within last 3 months or more than 3 months in the course of the disease
5. Are not simultaneously participating in another study which includes an investigational drug or procedure at study entry
6. Have been fully informed and given their written consent for use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population consists of adult patients with type 2 diabetes mellitus treated in outpatient setting by specialists.
Sampling Method: Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (50):
- Italy (50):
  - Research site, Acquaviva delle Fonti
  - Research site, Anzio
  - Research site, Bassano del Grappa
  - Research site, Bologna
  - Research site, Brindisi
  - Research site, Cagliari
  - Research site, Campi Salentina
  - Research site, Casarano
  - Research site, Caserta
  - Research site, Cesena
  - Research site, Chieri
  - Research site, Cisternino
  - Research site, Copertino
  - Research site, Cremona
  - Research site, Distretto Vittoria
  - Research site, Fermo
  - Research site, Ferrara
  - Research site, Fidenza
  - Research site, Florence
  - Research site, Forlì
  - Research site, Genova
  - Research site, Germaneto
  - Research site, Lecce
  - Research site, Livorno
  - Research site, Lucca
  - Research site, Manfredonia (Le)
  - Research site, Mariano Comense
  - Research site, Messina
  - Research site, Milan
  - Research site, Monza
  - Research site, Napoli
  - Research site, Novara
  - Research site, Olbia
  - Research site, Palermo
  - Research site, Palmi
  - Research site, Parma
  - Research site, Pavia
  - Research site, Pisa
  - Research site, Potenza
  - Research site, Rimini
  - Research site, Roma
  - Research site, Rossano Scalo
  - Research site, Salerno
  - Research site, San Giovanni Rotondo
  - Research site, Schio
  - Research site, Sesto San Giovanni
  - Research site, Siena
  - Research site, Treviso
  - Research site, Trieste
  - Research site, Varese

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six patients were not assigned to any cohort because the type of treatment taken was not reported.
Groups:
- Exenatide: The targeted population consists of adult patients with type 2 Diabetes Mellitus unable to achieve the desired level of glycemic control while using oral anti-hyperglycemic agents and who initiate treatment with exenatide.
  exenatide : subcutaneous injection, 5mcg or 10mcg, twice a day
- Basal Insulin: The targeted population consists of adult patients with type 2 Diabetes Mellitus unable to achieve the desired level of glycemic control while using oral anti-hyperglycemic agents and who initiate treatment with basal insulin.
  basal insulin : subcutaneous injection, dosing according to physician's clinical judgment
Period: Overall Study
Arm/Group | Exenatide | Basal Insulin
Started | 444 | 438
Completed | 377 | 371
Not Completed | 67 | 67
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 18 | 34
Not completed — entry criteria not met | 4 | 3
Not completed — Withdrawal by Subject | 35 | 23
Not completed — lack of glycemic control | 2 | 1
Not completed — lack of compliance | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Basal Insulin | Total
Number analyzed (Participants) | 444 | 438 | 882
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.65) | 65.9 (9.62) | 62.5 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 191 | 389
  Male | 246 | 247 | 493
Weight [Mean (Standard Deviation); unit: kg] | 97.5 (21.39) | 79.5 (15.82) | 88.6 (20.91)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] | 8.7 (1.34) | 9.2 (1.40) | 8.9 (1.39)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved Glycemic Target of HbA1c ≤ 7.0% With Minimal Weight Gain (≤ 1 Kg) at Month 12.
Description: Percentage of patients who achieved glycemic target of HbA1c ≤ 7.0% with minimal weight gain (≤ 1 Kg) at month 12.
Time Frame: Baseline, Month 12
Population: All patients who provided consent to release information and who fulfill the study entry criteria were included in the analyses.
  Patients were assigned to the exenatide BID or insulin cohort based on their initial injectable treatment started at baseline, and analyses were conducted irrespective of later treatment changes.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 397 | 405
percentage of patients | 35.0 [30.32 to 39.93] | 15.8 [12.39 to 19.73]

2. Secondary Outcome: Changes in HbA1c From Baseline to Month 12
Description: Changes in HbA1c from Baseline to Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 379 | 364
percent | -1.1 (1.40) | -1.4 (1.49)

3. Secondary Outcome: Changes in Fasting Blood Glucose From Baseline to Month 12
Description: Changes in Fasting Blood Glucose From Baseline to Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 303 | 287
mg/dL | -26.7 (57.05) | -51.4 (64.53)

4. Secondary Outcome: Percentage of Patients With HbA1c Reduction From Baseline >= 1.0% at Month 12
Description: Percentage of Patients with HbA1c Reduction from Baseline >= 1.0% at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 397 | 405
percentage of patients | 49.4 | 51.1

5. Secondary Outcome: Percentage of Patients Achieving HbA1c Concentration <=7.0% at Month 12
Description: Percentage of Patients Achieving HbA1c Concentration <=7.0% at Month 12
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 397 | 405
percentage of patients | 39.0 | 22.2

6. Secondary Outcome: Percentage of Patients Achieving HbA1c Concentration <6.5% at Month 12
Description: Percentage of Patients Achieving HbA1c Concentration <6.5% at Month 12
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 397 | 405
percentage of patients | 13.1 | 4.9

7. Secondary Outcome: Changes in Weight From Baseline to Month 12
Description: Changes in Weight From Baseline to Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 377 | 366
kg | -3.9 (5.92) | 0.2 (4.78)

8. Secondary Outcome: Percentage of Patients Achieving a Weight Decrease >=3% Between Baseline and Month 12
Description: Percentage of Patients Achieving a Weight Decrease >=3% between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
percentage of patients | 43.0 | 17.6

9. Secondary Outcome: Percentage of Patients Achieving a Weight Decrease >=5% Between Baseline and Month 12
Description: Percentage of Patients Achieving a Weight Decrease >=5% between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
percentage of patients | 29.7 | 10.7

10. Secondary Outcome: Changes in Fasting Total Cholesterol Between Baseline and Month 12
Description: Changes in Fasting Total Cholesterol Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 249 | 225
mg/dL | -6.0 (36.22) | -7.5 (43.58)

11. Secondary Outcome: Changes in Fasting HDL Between Baseline and Month 12
Description: Changes in Fasting HDL Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 226 | 203
mg/dL | 1.3 (10.12) | 0.2 (10.18)

12. Secondary Outcome: Changes in Fasting LDL Between Baseline and Month 12
Description: Changes in Fasting LDL Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 164 | 138
mg/dL | -4.6 (30.79) | -4.5 (38.35)

13. Secondary Outcome: Changes in Fasting Triglycerides Between Baseline and Month 12
Description: Changes in Fasting Triglycerides Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 240 | 226
mg/dL | -16.5 (115.27) | -30.2 (108.15)

14. Secondary Outcome: Changes in Diastolic Blood Pressure Between Baseline and Month 12
Description: Changes in Diastolic Blood Pressure Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 369 | 360
mmHg | -2.4 (10.40) | 0.2 (10.20)

15. Secondary Outcome: Changes in Systolic Blood Pressure Between Baseline and Month 12
Description: Changes in Systolic Blood Pressure Between Baseline and Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 369 | 360
mmHg | -4.6 (18.74) | -1.0 (17.56)

16. Secondary Outcome: Percentage of Patients With Hypoglycemia Episodes Between Baseline and Month 12
Description: Percentage of patients with Hypoglycemia Episodes Between Baseline and Month 12.
  All episodes consistent with hypoglycemia with or without a confirmatory blood glucose reading were collected.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
percentage of patients | 3.6 | 8.2

17. Secondary Outcome: Factors of Gender, Baseline Presence of Medical Conditions, and Previous Gastrointestinal Symptoms Associated With Treatment Choice at Baseline
Description: Number of patients per arm who were evaluated in 3 factors at baseline (gender, presence of medical conditions, and previous gastrointestinal symptoms) were analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor.
Time Frame: baseline
Population: All patients consented to release information; fulfilled study entry criteria. Analyses conducted on baseline arm assignment, irrespective of later treatment changes. Only those assigned to an arm were included. Missing values for numeric covariates replaced with means; categorical ones, with modes.
Measure: Number; unit: participants
Groups:
- Exenatide: The targeted population consists of adult patients with type 2 Diabetes Mellitus unable to achieve the desired level of glycemic control while using oral anti-hyperglycemic agents and who initiate treatment with exenatide. Exenatide subcutaneous injection, 5mcg or 10mcg, twice a day.
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
participants
  Male Gender | 246 [0.62 to 1.46] | 247
  Female Gender | 198 | 191
  Medical conditions present | 371 [0.74 to 1.76] | 363
  No medical conditions | 73 | 75
  Previous gastrointestinal symptoms present | 8 [0.43 to 3.42] | 11
  No gastrointestinal symptoms | 436 | 427
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if Baseline Gender (Male vs. Female), was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.831, Regression, Logistic; If several variables had Spearman's rho > 0.4 (for continuous) and Cramer's V > 0.4 (for categorical covariates), only one was left in the model; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.62 to 1.46]
Statistical Analysis 2: Comparison: Exenatide; Logistic regression analysis was used to find factors associated with treatment choice at baseline. Covariates with more than 30% observations missing are omitted in this analysis. Weight was removed (high correlation with BMI) and also fasting blood glucose (lab value) was removed (high correlation with HbA1c). Missing values for remaining numeric covariates were replaced with means, and for categorical ones-with modes; Test type: Superiority or Other; p = 0.554, Regression, Logistic — Baseline Medical conditions (yes vs. no); Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.74 to 1.76]
Statistical Analysis 3: Comparison: Exenatide; [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; p = 0.714, Regression, Logistic — Baseline gastrointestinal symptoms (yes vs. no); Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.43 to 3.42]

18. Secondary Outcome: Factor of 1 Percent (%) Higher Baseline HbA1c Associated With Treatment Choice at Baseline
Description: Factor of 1% higher baseline HbA1c (from most recent HbA1c) was analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. HbA1c was measured as a percent of normal (%).
Time Frame: baseline
Population: Full analysis set (FAS) population: all patients who provided consent to release information and who fulfilled the study entry criteria.
  FAS=444, however 1 patient in the exenatide arm was missing data for the most recent HbA1c at baseline so n=443.
Measure: Mean (Standard Deviation); unit: Percentage of normal
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 443 | 438
Percentage of normal | 8.7 (1.34) | 9.2 (1.40)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if Baseline HbA1c was 1% more, was it associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.60 to 0.78]

19. Secondary Outcome: Factor of Longer Duration of Diabetes Associated With Treatment Choice at Baseline
Description: The Factor of longer duration of diabetes at baseline (diagnosed 1 year longer) was analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. Duration of diabetes was measured in years since the date of diabetes diagnosis.
Time Frame: baseline
Population: Full analysis set (FAS) population: all patients who provided consent to release information and who fulfilled the study entry criteria.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
years | 9.0 (7.03) | 12.4 (8.29)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if longer duration of diabetes was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.055, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.96 to 1.00]

20. Secondary Outcome: Factor of Older Age Associated With Treatment Choice at Baseline
Description: Older age (1 year older) was analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. Age was measured in years.
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 438
years | 59.2 (9.65) | 65.9 (9.62)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if older age (1 year older), was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.95 to 0.99]

21. Secondary Outcome: Factor of Higher Body Mass Index (BMI) Associated With Treatment Choice at Baseline
Description: Factor of higher body mass index (BMI) (1 kilogram per meter squared (kg/m^2) higher) was analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. BMI measured as kg/m^2.
Time Frame: baseline
Population: Full analysis set (FAS) population: all patients who provided consent to release information and who fulfilled the study entry criteria.
  FAS for basal insulin arm=438 but one patient did not have data in this arm so n=437.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 437
kg/m^2 | 35.4 (6.83) | 29.4 (5.12)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if higher BMI (1 kg/m^2 higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.15 to 1.23]

22. Secondary Outcome: Factor of Greater Height Associated With Treatment Choice at Baseline
Description: Factor of greater height (1 centimeter higher) was analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. Height was measured in centimeters (cm) .
Time Frame: baseline
Population: Full analysis set (FAS) population: all patients who provided consent to release information and who fulfilled the study entry criteria.
  FAS for basal insulin arm=438 but one patient did not provide height data so n=437.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 444 | 437
cm | 165.8 (9.56) | 164.4 (9.10)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if greater height (1 cm higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.026, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [1.00 to 1.05]

23. Secondary Outcome: Factors of Higher Creatinine, Higher Fasting High Density Lipoprotein (HDL) Cholesterol, Higher Fasting Cholesterol, and Higher Fasting Triglycerides Which Were Associated With Treatment Choice at Baseline
Description: Factors of higher creatinine: 1 milligram per deciliter higher (mg/dL) and higher fasting lipids (HDL cholesterol: 1 mg/dL higher; total cholesterol: 1 mg/dL higher; triglycerides: 1 mg/dL higher) were analyzed for association with treatment choice at baseline. A total of 12 factors were evaluated. A multivariate logistic regression model using the full analysis set (FAS) population was performed for each of the factors to determine if exenatide treatment was more likely to be initiated in the presence of the specific factor. Creatinine and fasting lipids were measured in milligrams per deciliter (mg/dL).
Time Frame: baseline
Population: Full analysis set (FAS) population: all patients who provided consent to release information and who fulfilled the study entry criteria. FASS=444 and 438 in each arm respectively but the number of patients with creatinine and fasting lipids data at baseline varied. N is presented with each category.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Basal Insulin
Number analyzed (Participants) | 368 | 360
mg/dL
  Creatinine (N=324, 333) | 0.9 (0.24) | 1.0 (0.39)
  HDL (N=335, 326) | 44.7 (12.82) | 46.9 (12.31)
  Total Cholesterol (N=368, 355) | 181.1 (40.00) | 182.7 (41.79)
  Triglycerides (N=364, 360) | 177.5 (112.57) | 173.6 (104.24)
Statistical Analysis 1: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if higher baseline creatinine (1mg/dL higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.007, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.18 to 0.77]
Statistical Analysis 2: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if higher baseline fasting HDL cholesterol (1mg/dL higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.094, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.97 to 1.00]
Statistical Analysis 3: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if higher baseline fasting total cholesterol (1mg/dL higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.259, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [1.00 to 1.01]
Statistical Analysis 4: Comparison: Exenatide vs Basal Insulin; Logistic regression analysis was used to determine if higher baseline fasting triglycerides (1mg/dL higher) was associated with treatment choice at baseline. Odds ratios were determined and if the odds ratio was greater than 1, it indicated it is more likely to initiate exenatide treatment. Covariates with more than 30% observations missing were omitted in this analysis. Missing values for remaining numeric covariates were replaced with means, and for categorical ones - with modes; Test type: Superiority or Other; p = 0.123, Regression, Logistic; [statistical method as in outcome 17, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [1.00 to 1.00]

ADVERSE EVENTS:
Arm/Group | Exenatide | Basal Insulin
Serious Adverse Events (participants affected / at risk) | 11/444 | 10/438
Other Adverse Events (participants affected / at risk) | 19/444 | 9/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=444) | Basal Insulin (N=438)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (2)
Coma hepatic (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=444) | Basal Insulin (N=438)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No